CLINICAL TRIAL: NCT04031222
Title: Mechanisms of Inflammation, Immunity, Islet Cell and Intestinal Hormone Changes in Youth at Risk for Diabetes (MI4D)
Brief Title: Mechanisms of Inflammation, Immunity, Islet Cell and Intestinal Hormone Changes in Youth at Risk for Diabetes
Acronym: MI4D
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Toronto (Other); University of Guelph (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Staff Endocrinologist, Division Head, Endrocrinology, The Hospital for Sick Children
Other Study IDs: 1000055159
Record Dates: First submitted 2019-07-10; First posted 2019-07-24 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Obesity; PreDiabetes; Adolescent Obesity; Inflammation; Metabolic Problems; Insulin Resistance; Gut Microbiome; Immunity; Beta Cell Dysfunction; Gut Hormones
MeSH Terms: conditions — Obesity; Prediabetic State; Pediatric Obesity; Inflammation; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to assess the role of inflammation in insulin resistant conditions (i.e., obesity and pre-diabetes) and the subsequent development of disease, such as type 2 diabetes (T2D) and cardiovascular disease (CVD), in the adolescent population.

DETAILED DESCRIPTION:
This study proposes to characterize inflammatory biomarkers, insulin resistance and fecal microbiome composition in obese/pre-diabetic adolescents after glucose ingestion, followed by an oral fat tolerance test on a separate visit. Lipoprotein abnormalities and intestinal biomarkers, post-lipid ingestion, will also be evaluated. The primary aim is to assess the role of inflammation in insulin resistant conditions (i.e., obesity and pre-diabetes) and the subsequent development of disease, such as type 2 diabetes (T2D) and cardiovascular disease (CVD), in the adolescent population.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 12 - 18 years old with obesity (defined as body mass index (BMI) >97th percentile based on their age- and sex-specific World Health Organization growth chart)

Exclusion Criteria:

1. Known type 2 diabetes
2. Diabetes secondary to medication or surgery
3. Antibodies suggestive of type 1 diabetes
4. Pregnancy
5. Were born by C-section
6. Developmental delay precluding assent/consent
7. Acute illness within the past 3 days (chills, fever, vomiting > 1x, or diarrhea > 3x)
8. Taking medications that influence glucose (e.g., steroids, metformin) or lipids (e.g., statins)
9. Have taken prescribed medicine/antibiotics in the three months prior to clinic or study visit
10. Significant chronic illness (e.g., Cushing's Disease, Craniopharyngioma, Hypothalamic Obesity, etc.)
11. Lactose intolerance and/or milk allergy (Study Visit Day 2 Only)
12. Bariatric surgery

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with obesity
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Whole body insulin sensitivity index | Through study completion, an average of 2 years.
  Multiple measurements from a 2-hour oral glucose tolerance will be aggregated to arrive at one reported value (ie., insulin in uU/mL units and glucose values in mg/dL units which are measured at baseline, 30 min, 60 min, 90 min, and 120 min during the oral glucose tolerance test will be combined to calculate whole body insulin sensitivity index). There is no unit of measure for whole body insulin sensitivity index. Whole body insulin sensitivity index will be calculated using the following equation: whole body insulin sensitivity index = 10,000 / √ [(fasting glucose x fasting insulin) x (mean glucose x mean insulin)].
Microbiome Composition | Through study completion, an average of 3 years.
  We will perform microbiome 16S ribosomal ribonucleic acid (rRNA) sequencing in fecal samples from study participants.
Inflammatory markers | Through study completion, an average of 3 years.
  Cytokines will be measured in plasma and fecal water with Bio-PlexTM arrays providing biomarkers of type 1 diabetes and/or type 2 diabetes progression. As indices of gut microbial translocation, serum lipopolysaccharides (LPS), macrophage secreted cluster of differentiation 14 (CD14) that binds LPS and LPS binding protein (LBP) will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Jill K Hamilton, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada